CLINICAL TRIAL: NCT00713609
Title: A Multi-center, Randomized, Double-blind, Vehicle-Controlled, Phase 2 Study of the Safety and Efficacy of Benzoyl Peroxide/Clindamycin Gel and Tazarotene Cream When Used in Combination in the Treatment of Acne Vulgaris
Brief Title: Safety and Efficacy Study of Clindamycin/Benzoyl Peroxide/Tazarotene Cream in Subjects With Acne
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114570
Record Dates: First submitted 2008-07-07; First posted 2008-07-11 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Acne Vulgaris
Keywords: Acne; Acne Vulgaris; Pimples
MeSH Terms: conditions — Acne Vulgaris | interventions — clindamycin phosphate benzoyl peroxide combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): Benzoyl peroxide/clindamycin gel + tazarotene cream
  Interventions: Drug: Benzoyl peroxide gel; Drug: Clindamycin gel; Drug: Tazarotene cream
- 2 (Active Comparator): Benzoyl peroxide/clindamycin gel + vehicle cream
  Interventions: Drug: Benzoyl peroxide gel; Drug: Clindamycin gel; Drug: Vehicle cream
- 3 (Active Comparator): Benzoyl peroxide gel + tazarotene cream
  Interventions: Drug: Benzoyl peroxide gel; Drug: Tazarotene cream
- 4 (Active Comparator): Clindamycin gel + tazarotene cream
  Interventions: Drug: Clindamycin gel; Drug: Tazarotene cream
- 5 (Active Comparator): Vehicle gel+ tazarotene cream
  Interventions: Drug: Tazarotene cream; Drug: Vehicle gel
- 6 (Placebo Comparator): Vehicle gel + vehicle cream
  Interventions: Drug: Vehicle gel; Drug: Vehicle cream

INTERVENTIONS:
Drug: Benzoyl peroxide gel — 5% benzoyl peroxide in a gel applied topically once a day
  Arms: 1; 2; 3
Drug: Clindamycin gel — 1% clindamycin phosphate applied topically once a day
  Arms: 1; 2; 4
Drug: Tazarotene cream — 0.1 % tazarotene in a cream applied topically once a day
  Arms: 1; 3; 4; 5
Drug: Vehicle gel — Vehicle gel is an identical gel without the active ingredients
  Arms: 5; 6
Drug: Vehicle cream — Vehicle cream is an identical cream without the active ingredients
  Arms: 2; 6

SUMMARY:
Benzoyl peroxide, clindamycin and tazarotene are known to be effective treatment alternative for acne vulgaris. The purpose of this study is to assess the safety and efficacy of a combination product including these actives for the treatment of acne vulgaris.

You may be suitable to take part in this study because you have acne vulgaris on your face. Acne vulgaris usually affects the face, but it can also affect the skin on the chest, arms, legs, and back.

DETAILED DESCRIPTION:
The study subjects must have acne vulgaris and will apply study drug to their face for 12 weeks.

Study visits will occur at baseline (day 1) and at weeks 2, 4, 8, and 12. Subjects will be assessed at every visit to determine how the study drug is working. Safety will be assessed by evaluation of adverse events (AEs), vital signs, physical examinations, and withdrawals from the study.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria: Subjects must be males or females 12 to 45 years of age.
* Subjects must have acne on their face.
* Female subjects of childbearing potential must have a negative pregnancy test. If sexually active, one medically acceptable forms of contraception must be practiced from baseline to the last study visit.
* Subjects must have the ability and willingness to follow all study procedures, attend all scheduled visits, and successfully complete the study.
* Subjects must be capable of understanding and willing to provide signed and dated written voluntary informed consent (and any local or national authorization requirements).
* Subjects must be able to complete the study and to comply with study instructions.

Exclusion Criteria:

* Subjects who are pregnant, trying to become pregnant, or breast-feeding.
* Subjects with conditions that may influence the safety and or efficacy assessments of the study including, but not limited to: regional enteritis or inflammatory bowel disease, lupus, dermatomyositis, rosacea, seborrheic dermatitis, beard folliculitis, or perioral dermatitis, subject who are immunocompromised or have had any major illness within 30 days before the screening examination
* History of known or suspected intolerance including any known hypersensitivity or previous allergic reaction to any of the ingredients of the study products
* Subjects who have used topical antibiotics or topical steroids on the face, facial procedures, or any investigational therapy within the past 4 weeks or systemic retinoids within the past 6 months.
* Subjects who have any other disease or condition, or are using any medication, that in the judgment of the investigator would put the subject at unacceptable risk for participation in the study.
* Other exclusion criteria may apply.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 591 (Actual)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- United States (16):
  - Dermatology Research of Arkansas, Little Rock, Arkansas
  - Center for Dermatology Cosmetic and Laser Surgery, Fremont, California
  - Center for Dermatology and Laser Surgery, Sacramento, California
  - Boulder Medical Center, P.C., Boulder, Colorado
  - Dermatology Associates Research, Coral Gables, Florida
  - MedaPhase, Inc., Newnan, Georgia
  - Callender Center for Clinical Research, Mitchellville, Maryland
  - Grekin Skin Institute, Warren, Michigan
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Dermatology Consulting Services, High Point, North Carolina
  - MS Hershey Medical Center, Hershey, Pennsylvania
  - Rivergate Dermatology & Skin Care Center, Goodlettsville, Tennessee
  - The Skin Wellness Center, PC, Knoxville, Tennessee
  - Dermatology Treatment & Research Center, Dallas, Texas
  - Suzanne Bruce and Associates, PA, Houston, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this multi-center, double-blind, vehicle controlled study, participants were assigned to one of the six treatment groups in a 2:2:2:2:2:1 ratio for 12 weeks.
Pre-assignment Details: Participants with facial acne vulgaris, 12 to 45 years of age were enrolled in this study. A total of 596 participants were randomized and 587 participants received study product.
Groups:
- Benzoyl Peroxide/Clindamycin + Tazarotene: Participants applied the study product (Benzoyl peroxide/Clindamycin + Tazarotene) to the face once daily in the evening up to 12 weeks. Two actuations of test product (approximately 0.6 grams [g] of the combined product in an approximate 1:1 ratio) were dispensed into the participant's palm and mixed. A thin film was then applied to the entire face
- Benzoyl Peroxide/Clindamycin + Vehicle Cream: Participants applied the study product (Benzoyl peroxide/Clindamycin + vehicle cream with identical ingredients as Tazarotene) to the face once daily in the evening up to 12 weeks. Two actuations of test product (approximately 0.6 g of the combined product in an approximate 1:1 ratio) were dispensed into the participant's palm and mixed. A thin film was then applied to the entire face.
- Benzoyl Peroxide Gel + Tazarotene: Participants applied the study product (Benzoyl peroxide gel + Tazarotene) to the face once daily in the evening up to 12 weeks. Two actuations of test product (approximately 0.6 g of the combined product in an approximate 1:1 ratio) were dispensed into the participant's palm and mixed. A thin film was then applied to the entire face.
- Clindamycin Gel + Tazarotene: Participants applied the study product (Clindamycin gel + Tazarotene) to the face once daily in the evening up to 12 weeks. Two actuations of test product (approximately 0.6 g of the combined product in an approximate 1:1 ratio) were dispensed into the participant's palm and mixed. A thin film was then applied to the entire face.
- Vehicle Gel + Tazarotene: Participants applied the study product (Vehicle gel with identical ingredients as Benzoyl peroxide/Clindamycin + Tazarotene) to the face once daily in the evening up to 12 weeks. Two actuations of test product (approximately 0.6 g of the combined product in an approximate 1:1 ratio) were dispensed into the participant's palm and mixed. A thin film was then applied to the entire face.
- Vehicle Gel + Vehicle Cream: Participants applied the study product (Vehicle gel with identical ingredients as Benzoyl peroxide/Clindamycin+ vehicle cream with identical ingredients as Tazarotene) to the face once daily in the evening up to 12 weeks. Two actuations of test product (approximately 0.6 g of the combined product in an approximate 1:1 ratio) were dispensed into the participant's palm and mixed. A thin film was then applied to the entire face.
Period: Overall Study
Arm/Group | Benzoyl Peroxide/Clindamycin + Tazarotene | Benzoyl Peroxide/Clindamycin + Vehicle Cream | Benzoyl Peroxide Gel + Tazarotene | Clindamycin Gel + Tazarotene | Vehicle Gel + Tazarotene | Vehicle Gel + Vehicle Cream
Started | 106 | 105 | 107 | 108 | 106 | 55
Completed | 85 | 90 | 92 | 99 | 87 | 47
Not Completed | 21 | 15 | 15 | 9 | 19 | 8
Not completed — Adverse Event | 2 | 0 | 2 | 2 | 3 | 1
Not completed — Lost to Follow-up | 5 | 7 | 5 | 5 | 7 | 0
Not completed — Lack of Efficacy | 1 | 3 | 0 | 0 | 1 | 0
Not completed — Non-Compliance with Study Treatment | 1 | 1 | 2 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 6 | 1 | 5 | 1 | 5 | 7
Not completed — Protocol Violation | 6 | 3 | 1 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Benzoyl Peroxide/Clindamycin + Tazarotene | Benzoyl Peroxide/Clindamycin + Vehicle Cream | Benzoyl Peroxide Gel + Tazarotene | Clindamycin Gel + Tazarotene | Vehicle Gel + Tazarotene | Vehicle Gel + Vehicle Cream | Total
Number analyzed (Participants) | 106 | 105 | 107 | 108 | 106 | 55 | 587
Age, Continuous [Mean (Standard Deviation); unit: Years] | 19.7 (6.6) | 19.7 (6.9) | 20.2 (7.3) | 19.2 (6.2) | 21.7 (8.4) | 19.8 (6.6) | 20.1 (7.1)
Gender [Count of Participants; unit: Participants]
  Female | 58 | 56 | 60 | 60 | 65 | 35 | 334
  Male | 48 | 49 | 47 | 48 | 41 | 20 | 253
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 8 | 14 | 5 | 6 | 9 | 5 | 47
  Black | 23 | 16 | 24 | 15 | 14 | 8 | 100
  Multiracial | 10 | 11 | 9 | 8 | 8 | 5 | 51
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 0 | 1 | 0 | 4
  White | 63 | 63 | 68 | 79 | 74 | 37 | 384

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Lesion Counts (Total, Inflammatory, and Non-inflammatory) From Baseline to Week 12
Description: The investigator or designee took count of inflammatory lesions (papules, pustules, nodules and cysts [only post-Baseline]) (ILC), noninflammatory lesions (open and closed comedones) (NILC) and total lesions (TLC) at Baseline, Weeks 2, 4, 8, and 12. Lesion counts were confined to the face. Each of 3 lesion counts (total, inflammatory and non-inflammatory) was analyzed using an analysis of covariance (ANCOVA) model with terms for treatment, center, Baseline value and treatment-by-center interaction. If the interaction was not significant at 0.1 level, this interaction was excluded in ANCOVA model. Day 1 (Visit 1) was defined as Baseline. Only participants available at specified timepoints were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to Week 12
Population: Intent-to-treat (ITT) Analysis Set: all randomized participants who received study product and reached Week 12.
Measure: Mean (Standard Deviation); unit: Lesion count
Arm/Group | Benzoyl Peroxide/Clindamycin + Tazarotene | Benzoyl Peroxide/Clindamycin + Vehicle Cream | Benzoyl Peroxide Gel + Tazarotene | Clindamycin Gel + Tazarotene | Vehicle Gel + Tazarotene | Vehicle Gel + Vehicle Cream
Number analyzed (Participants) | 106 | 105 | 107 | 107 | 106 | 55
Lesion count
  ILC, n=101, 103, 105, 105, 104, 52 | -16.8 (14.35) | -18.1 (14.45) | -18.9 (12.84) | -18.8 (11.49) | -14.5 (12.76) | -8.96 (12.63)
  NILC, n=101, 103, 105, 105, 104, 52 | -33.0 (23.94) | -24.9 (33.41) | -37.1 (29.70) | -37.5 (29.51) | -33.0 (25.89) | -18.9 (28.41)
  TLC, n=101, 103, 105, 105, 104, 52 | -49.8 (31.78) | -43.0 (42.24) | -56.0 (34.99) | -56.3 (35.42) | -47.6 (33.32) | -27.8 (35.06)
Statistical Analysis 1: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Benzoyl Peroxide/Clindamycin + Vehicle Cream; Test type: Superiority or Other; p = 0.692, ANCOVA — For ILC
Statistical Analysis 2: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Benzoyl Peroxide Gel + Tazarotene; Test type: Superiority or Other; p = 0.467, ANCOVA — For ILC
Statistical Analysis 3: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Clindamycin Gel + Tazarotene; Test type: Superiority or Other; p = 0.281, ANCOVA — For ILC
Statistical Analysis 4: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Vehicle Gel + Tazarotene; Test type: Superiority or Other; p = 0.075, ANCOVA — For ILC
Statistical Analysis 5: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Vehicle Gel + Vehicle Cream; Test type: Superiority or Other; p < 0.001, ANCOVA — For ILC
Statistical Analysis 6: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Benzoyl Peroxide/Clindamycin + Vehicle Cream; Test type: Superiority or Other; p < 0.001, ANCOVA — For NILC
Statistical Analysis 7: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Benzoyl Peroxide Gel + Tazarotene; Test type: Superiority or Other; p = 0.803, ANCOVA — For NILC
Statistical Analysis 8: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Clindamycin Gel + Tazarotene; Test type: Superiority or Other; p = 0.175, ANCOVA — For NILC
Statistical Analysis 9: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Vehicle Gel + Tazarotene; Test type: Superiority or Other; p = 0.552, ANCOVA — For NILC
Statistical Analysis 10: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Vehicle Gel + Vehicle Cream; Test type: Superiority or Other; p < 0.001, ANCOVA — For NILC
Statistical Analysis 11: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Benzoyl Peroxide/Clindamycin + Vehicle Cream; Test type: Superiority or Other; p = 0.006, ANCOVA — For TC
Statistical Analysis 12: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Benzoyl Peroxide Gel + Tazarotene; Test type: Superiority or Other; p = 0.618, ANCOVA — For TC
Statistical Analysis 13: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Clindamycin Gel + Tazarotene; Test type: Superiority or Other; p = 0.149, ANCOVA — For TC
Statistical Analysis 14: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Vehicle Gel + Tazarotene; Test type: Superiority or Other; p = 0.255, ANCOVA — For TC
Statistical Analysis 15: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Vehicle Gel + Vehicle Cream; Test type: Superiority or Other; p < 0.001, ANCOVA — For TC

2. Primary Outcome: Proportion of Participants With a Minimum 2-grade Improvement in the Investigator's Static Global Assessment (ISGA) Score From Baseline to Week 12
Description: An ISGA was obtained at Baseline and at Weeks 2, 4, 8, and 12. The scores range from 0-5 (0=clear skin with no inflammatory or non-inflammatory lesions; 5=very severe with many non-inflammatory and inflammatory lesions and more than a few nodular lesions (may have cystic lesions). The higher score indicates more severe. The area considered for the ISGA was confined to the face. When possible, the same efficacy assessor performed all ISGA assessments on the same participant at all visits. Day 1 (Visit 1) was defined as Baseline. Only participants available at specified time points were analyzed.
Time Frame: Baseline and up to Week 12
Population: ITT Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Benzoyl Peroxide/Clindamycin + Tazarotene | Benzoyl Peroxide/Clindamycin + Vehicle Cream | Benzoyl Peroxide Gel + Tazarotene | Clindamycin Gel + Tazarotene | Vehicle Gel + Tazarotene | Vehicle Gel + Vehicle Cream
Number analyzed (Participants) | 106 | 105 | 107 | 108 | 106 | 55
Percentage of participants | 22 | 22 | 31 | 36 | 20 | 5
Statistical Analysis 1: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Benzoyl Peroxide/Clindamycin + Vehicle Cream; Test type: Superiority or Other; p = 0.922, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Benzoyl Peroxide Gel + Tazarotene; Test type: Superiority or Other; p = 0.132, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Clindamycin Gel + Tazarotene; Test type: Superiority or Other; p = 0.020, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Vehicle Gel + Tazarotene; Test type: Superiority or Other; p = 0.706, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Vehicle Gel + Vehicle Cream; Test type: Superiority or Other; p = 0.009, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percent Change From Baseline to Week 12 in Each of 3 Lesion Counts (Total, Inflammatory, and Non-inflammatory)
Description: The investigator or designee took count of inflammatory lesions (papules, pustules, nodules and cysts) (ILC), noninflammatory lesions (open and closed comedones) (NILC) and total lesions (TLC) at Baseline, Weeks 2, 4, 8, and 12. Lesion counts were confined to the face. Each of 3 lesion counts (total, inflammatory and non-inflammatory) was analyzed using an analysis of covariance (ANCOVA) model with terms for treatment, center, Baseline value and treatment-by-center interaction. If the interaction was not significant at 0.1 level, this interaction was excluded in ANCOVA model. Day 1 (Visit 1) was defined as Baseline. Only participants available at specified timepoints were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to Week 12
Population: ITT Analysis Set
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Benzoyl Peroxide/Clindamycin + Tazarotene | Benzoyl Peroxide/Clindamycin + Vehicle Cream | Benzoyl Peroxide Gel + Tazarotene | Clindamycin Gel + Tazarotene | Vehicle Gel + Tazarotene | Vehicle Gel + Vehicle Cream
Number analyzed (Participants) | 106 | 105 | 107 | 108 | 106 | 55
Percent change
  ILC, n=101, 103, 105, 105, 104, 52 | -58.3 (45.57) | -62.4 (39.33) | -62.4 (34.83) | -65.7 (33.38) | -49.0 (40.90) | -33.5 (41.10)
  NILC, n=101, 103, 105, 105, 104, 52 | -58.0 (29.97) | -39.2 (51.29) | -60.6 (35.00) | -61.2 (31.60) | -53.1 (30.56) | -29.5 (44.05)
  TLC, n=101, 103, 105, 105, 104, 52 | -59.1 (29.96) | -47.9 (38.89) | -62.0 (29.42) | -63.4 (28.75) | -51.8 (29.18) | -31.5 (37.59)
Statistical Analysis 1: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Benzoyl Peroxide/Clindamycin + Vehicle Cream; Test type: Superiority or Other; p = 0.504, ANCOVA — For ILC
Statistical Analysis 2: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Benzoyl Peroxide Gel + Tazarotene; Test type: Superiority or Other; p = 0.504, ANCOVA — For ILC
Statistical Analysis 3: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Clindamycin Gel + Tazarotene; Test type: Superiority or Other; p = 0.177, ANCOVA — For ILC
Statistical Analysis 4: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Vehicle Gel + Tazarotene; Test type: Superiority or Other; p = 0.084, ANCOVA — For ILC
Statistical Analysis 5: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Vehicle Gel + Vehicle Cream; Test type: Superiority or Other; p < 0.001, ANCOVA — For ILC
Statistical Analysis 6: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Benzoyl Peroxide/Clindamycin + Vehicle Cream; Test type: Superiority or Other; p < 0.001, ANCOVA — For NILC
Statistical Analysis 7: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Benzoyl Peroxide Gel + Tazarotene; Test type: Superiority or Other; p = 0.776, ANCOVA — For NILC
Statistical Analysis 8: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Clindamycin Gel + Tazarotene; Test type: Superiority or Other; p = 0.465, ANCOVA — For NILC
Statistical Analysis 9: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Vehicle Gel + Tazarotene; Test type: Superiority or Other; p = 0.288, ANCOVA — For NILC
Statistical Analysis 10: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Vehicle Gel + Vehicle Cream; Test type: Superiority or Other; p < 0.001, ANCOVA — For NILC
Statistical Analysis 11: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Benzoyl Peroxide/Clindamycin + Vehicle Cream; Test type: Superiority or Other; p = 0.006, ANCOVA — For TC
Statistical Analysis 12: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Benzoyl Peroxide Gel + Tazarotene; Test type: Superiority or Other; p = 0.620, ANCOVA — For TC
Statistical Analysis 13: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Clindamycin Gel + Tazarotene; Test type: Superiority or Other; p = 0.291, ANCOVA — For TC
Statistical Analysis 14: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Vehicle Gel + Tazarotene; Test type: Superiority or Other; p = 0.085, ANCOVA — For TC
Statistical Analysis 15: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Vehicle Gel + Vehicle Cream; Test type: Superiority or Other; p < 0.001, ANCOVA — For TC

4. Secondary Outcome: Proportion of Participants With an ISGA Score of 0 or 1 at Week 12
Description: as for outcome 2
Time Frame: Week 12
Population: ITT Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Benzoyl Peroxide/Clindamycin + Tazarotene | Benzoyl Peroxide/Clindamycin + Vehicle Cream | Benzoyl Peroxide Gel + Tazarotene | Clindamycin Gel + Tazarotene | Vehicle Gel + Tazarotene | Vehicle Gel + Vehicle Cream
Number analyzed (Participants) | 106 | 105 | 107 | 108 | 106 | 55
Percentage of participants | 33 | 31 | 27 | 39 | 22 | 13
Statistical Analysis 1: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Benzoyl Peroxide/Clindamycin + Vehicle Cream; Test type: Superiority or Other; p = 0.652, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Benzoyl Peroxide Gel + Tazarotene; Test type: Superiority or Other; p = 0.279, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Clindamycin Gel + Tazarotene; Test type: Superiority or Other; p = 0.312, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Vehicle Gel + Tazarotene; Test type: Superiority or Other; p = 0.063, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Benzoyl Peroxide/Clindamycin + Tazarotene vs Vehicle Gel + Vehicle Cream; Test type: Superiority or Other; p = 0.005, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from Day 1 up to Day 89.
Description: SAEs and non-serious AEs were assessed in the ITT Analysis Set.
Arm/Group | Benzoyl Peroxide/Clindamycin + Tazarotene | Benzoyl Peroxide/Clindamycin + Vehicle Cream | Benzoyl Peroxide Gel + Tazarotene | Clindamycin Gel + Tazarotene | Vehicle Gel + Tazarotene | Vehicle Gel + Vehicle Cream
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/105 | 0/107 | 0/108 | 0/106 | 0/55
Other Adverse Events (participants affected / at risk) | 25/106 | 22/105 | 24/107 | 18/108 | 29/106 | 12/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Benzoyl Peroxide/Clindamycin + Tazarotene (N=106) | Benzoyl Peroxide/Clindamycin + Vehicle Cream (N=105) | Benzoyl Peroxide Gel + Tazarotene (N=107) | Clindamycin Gel + Tazarotene (N=108) | Vehicle Gel + Tazarotene (N=106) | Vehicle Gel + Vehicle Cream (N=55)
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lip blister (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tooth impacted (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Application site burn (General disorders) | 0 | 0 | 1 | 0 | 1 | 1
Application site dermatitis (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Application site discolouration (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Application site dryness (General disorders) | 1 | 0 | 1 | 1 | 1 | 1
Application site erythema (General disorders) | 1 | 0 | 2 | 1 | 0 | 1
Application site exfoliation (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Application site irritation (General disorders) | 1 | 0 | 3 | 4 | 2 | 0
Application site pain (General disorders) | 0 | 0 | 2 | 0 | 0 | 2
Application site pruritus (General disorders) | 0 | 0 | 0 | 0 | 2 | 1
Condition aggravated (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cyst (General disorders) | 0 | 1 | 0 | 1 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Allergy to arthropod bite (Immune system disorders) | 2 | 0 | 0 | 0 | 1 | 0
Allergy to metals (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Food allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Multiple allergies (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 3 | 3 | 5 | 4 | 3
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 2 | 0 | 1 | 2
Tinea pedis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 4 | 5 | 2 | 4 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Vaginitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Smear cervix abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1
Fibromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 0
Insomnia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 2 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Wisdom teeth removal (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.